CLINICAL TRIAL: NCT02374853
Title: Topical Use of Vancomycin in Reducing Sternal Wound Infection in Cardiac Surgery (SWI Trial)
Acronym: SWI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: the preliminary analysis of study result did not show significant benefit that was anticipate
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SWI-01-14
Record Dates: First submitted 2015-02-23; First posted 2015-03-02 (Estimated); Results first posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-08

CONDITIONS: INFECTION
MeSH Terms: conditions — Infections | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vancomycin (Experimental): During open heart surgery, patients will have a 4 x 8 inch piece of sterile gauze covering each side of the divided sternum. The gauze will be soaked in the following solution: 5 g vancomycin dissolved in 50 mL sterile water
  Interventions: Drug: Vancomycin
- Control (Placebo Comparator): During open heart surgery, patients will have a 4 x 8 inch piece of sterile gauze covering each side of the divided sternum. The gauze will be soaked in 50 mL sterile water. No Vancomycin
  Interventions: Other: No Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Topical prophylactic antibiotic
  Other Names: Vancomycin Hydrochloride
  Arms: Vancomycin
Other: No Vancomycin — Placebo: Sterile water. No Vancomycin.
  Other Names: Sterile water
  Arms: Control

SUMMARY:
The purpose of this research is to determine if using the antibiotic vancomycin as a preventative topical (on the surface of the skin) treatment during open-heart surgery will reduce the risk of developing a sternal wound infection.

DETAILED DESCRIPTION:
During open-heart surgery, an incision is made along the chest and the sternum (breastbone) is divided. The sternum is held open throughout the surgery so that the doctors can reach the heart. Sternal wound infection is an uncommon but serious complication of cardiac surgery that occurs when an infection develops at this site of entry. Sternal wound infections are associated with increased hospital stays, subsequent surgical procedures, and higher mortality rates.

The purpose of this research is to determine if using the antibiotic vancomycin as a preventative topical (on the surface of the skin) treatment during open-heart surgery will reduce the risk of developing a sternal wound infection. The results of this study could provide important information to guide new standards of practice in cardiac surgery. The ultimate goal of this research project is to improve patient care by reducing the number of sternal wound infections at our hospital.

ELIGIBILITY:
Inclusion Criteria:

* Able to sign Informed Consent and Release of Medical Information Form
* Age ≥ 18 years
* Undergoing cardiac surgery with complete sternotomy (including re-operations)

Exclusion Criteria:

* Evidence of active infection (any culture positive or blood positive infection)
* Undergoing organ transplantation
* Patients with known hypersensitivity to vancomycin
* Pregnant or nursing women
* Mental impairment or other conditions that may not allow participant to understand the nature, significance, and scope of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1037 (Actual)
Dates: Start 2015-03; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abbas Khani-Hanjani, MD, Principal Investigator — University of Alberta

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vancomycin | Control
Started | 517 | 520
Completed | 512 | 509
Not Completed | 5 | 11
Not completed — Surgery Cancelled | 5 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vancomycin | Control | Total
Number analyzed (Participants) | 512 | 509 | 1021
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.61 (12.77) | 62.71 (13.49) | 63.16 (13.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 109 | 225
  Male | 396 | 400 | 796
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 512 | 509 | 1021
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg^m2] | 29.9 (5.8) | 30.1 (5.7) | 30.0 (5.8)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m2] | 2.1 (0.3) | 2.1 (0.3) | 2.1 (0.3)
Diabetes Mellitus [Count of Participants; unit: Participants] | 167 | 157 | 324

OUTCOME MEASURES:

1. Primary Outcome: Number of Sternal Wound Infections
Description: The number of sternal wound infections at 3 months postoperative. This includes superficial incisional, deep incisional, and organ/space surgical site infections.
Time Frame: 3 months postoperative
Measure: Number; unit: number of infections
Arm/Group | Vancomycin | Control
Number analyzed (Participants) | 512 | 509
number of infections | 14 | 21
Statistical Analysis 1: Comparison: Vancomycin vs Control; Test type: Superiority; p = 0.23, Fisher Exact

2. Secondary Outcome: Number of Sternal Wound Infections
Description: The number of sternal wound infections at 1 year postoperative. This includes superficial incisional, deep incisional, and organ/space surgical site infections.
Time Frame: 1 year postoperative
Measure: Number; unit: number of infections
Arm/Group | Vancomycin | Control
Number analyzed (Participants) | 512 | 509
number of infections | 15 | 22
Statistical Analysis 1: Comparison: Vancomycin vs Control; Test type: Superiority; p = 0.25, Fisher Exact

3. Secondary Outcome: Hospitalization
Description: Duration of index hospitalization and subsequent re-admissions due to sternal wound infection.
Time Frame: 1 year postoperative
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Vancomycin | Control
Number analyzed (Participants) | 512 | 509
days | 9.4 (9.0) | 8.7 (7.0)
Statistical Analysis 1: Comparison: Vancomycin; Test type: Superiority; p = .054, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Participants With Use of Prophylactic Antibiotics
Description: Number of participants with use of prophylactic antibiotics before surgery
Time Frame: Assessed before surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin | Control
Number analyzed (Participants) | 512 | 509
Participants | 512 | 509

5. Secondary Outcome: Cost Analysis for Sternal Wound Infection Treatment
Description: Cost analysis for sternal wound infection treatment post-operatively
Time Frame: 1 year postoperative
Population: Data were not collected.
Arm/Group | Vancomycin | Control
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Adverse Events
Description: Adverse events during study participation
Time Frame: 1 year postoperative
Measure: Number; unit: number of adverse events
Arm/Group | Vancomycin | Control
Number analyzed (Participants) | 512 | 509
number of adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: Post-operatively, 3 months and 1 year.
Arm/Group | Vancomycin | Control
All-Cause Mortality (participants affected / at risk) | 0/512 | 0/509
Serious Adverse Events (participants affected / at risk) | 0/512 | 0/509
Other Adverse Events (participants affected / at risk) | 0/512 | 0/509

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT02374853/Prot_SAP_000.pdf